CLINICAL TRIAL: NCT00989274
Title: Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of the Vaccine Against Pandemic Influenza A/H1N1 Produced by Sanofi
Brief Title: Clinical Trial to Evaluate the Immunogenicity and Safety of the Vaccine Against Influenza A/H1N1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Late approval by the Secretariat of Health, and expiration of vaccine
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Laboratorios de Biologicos y Reactivos de México, S.A. de C.V. (Other)
Responsible Party: Principal Investigator, Ma. de Lourdes Garcia Garcia, Director of the Center of Research in Infectious Diseases, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CI:863, No. 777
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Immunology; Immunogenicity; Reactogenicity; Safety; Influenza vaccine; Immune response; Adverse effects
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine Sanofi A(H1N1) 15 ug & trivalent (Active Comparator): 120 participants selected by random
  Interventions: Biological: Vaccine Sanofi A(H1N1) 15 ug & trivalent
- Vaccine Sanofi (H1N1) 15 ug.nonadyuvante (Active Comparator): 120 participants selected in random form
  Interventions: Biological: Vaccine Sanofi (H1N1) 15 ug.nonadyuvante
- Vaccine Sanofi A(H1N1) 7.5 ug (Active Comparator): 120 participants selected in random form
  Interventions: Biological: Vaccine Sanofi A(H1N1) 7.5 ug

INTERVENTIONS:
Biological: Vaccine Sanofi A(H1N1) 15 ug & trivalent — Grup 1: day 0: Vaccine trivalent (A/Brisbane/59/2007 (H1N1)-like virus, A/Brisbane/10/2007 (H3N2)-like virus, and B/Brisbane/60/2008-like virus) Vaccine Sanofi A(H1N1) administrated 15 ug. (nonadjuvant); day 28 Vaccine Sanofi A(H1N1) administrated a 15 ug. (nonadjuvant);
  Other Names: Vaccine Sanofi A(H1N1)
  Arms: Vaccine Sanofi A(H1N1) 15 ug & trivalent
Biological: Vaccine Sanofi (H1N1) 15 ug.nonadyuvante — Grup 2: Day 0: Vaccine trivalent(A/Brisbane/59/2007 (H1N1)-like virus, A/Brisbane/10/2007 (H3N2)-like virus, y B/Brisbane/60/2008-like virus); Day 28 Vaccine Sanofi A(H1N1) administrated a 15 ug. (nonadjuvant); day 56; Vaccine Sanofi A(H1N1) administrated a 15 ug. (nonadjuvant)
  Other Names: Vaccine Sanofi A(H1N1)
  Arms: Vaccine Sanofi (H1N1) 15 ug.nonadyuvante
Biological: Vaccine Sanofi A(H1N1) 7.5 ug — Grup 3: day 0: day 28 Vaccine Sanofi A(H1N1) administrated a 7.5 ug (non adjuvant); day 56; Vaccine Sanofi A(H1N1) administrated a 7.5 ug (nonadjuvant).
  Other Names: Vaccine Sanofi A(H1N1)
  Arms: Vaccine Sanofi A(H1N1) 7.5 ug

SUMMARY:
In agreement with the World Organization of the Health (WHO), during the annual epidemics of influenza they become infected between 10-20 % of the total population, appearing from a feverish disease up to leading to the hospitalization and in some cases to the death. To unpredictable intervals and due to the nature of the virus, this one can acquire new genes of others virus of the influenza that they concern birds or porks, of it it turns out to be a new virus with a completely new subtype of IT (HE,SHE) HAS and NA, and if this one is transmitted efficiently of person-to-person can cause a pandemic.

This phenomenon has been the one that has given place to the appearance of a new causative virus of the outbreak of influenza humanizes in Mexico (A/México/2009 (H1N1)), and in agreement to official Mexican numbers(figures), until August 13 there have been brought(reported) a whole of 18,861 cases and 163 deaths. The measure of the most effective control against the influenza constitutes it the vaccine, by what study becomes imperative to possess (to rely on) a vaccine against the new virus To (H1N1) East is relevant, due to the level of response of alert to a level 6 (pandemic) that has passed the World Organization of the Health (WHO).

DETAILED DESCRIPTION:
The originality of the study is based the fact that the study will be a clinical test(essay) phase the IInd for this new vaccine. Additional it will allow to obtain information in relation to the immunity crossed between(among) pandemic vaccines and seasonal vaccines. Equally it will allow to obtain evidence on the impact of the possible protection of the seasonal vaccine that is in use in the routine programs of vaccination in opposition to the virus of the influenza To (H1N1sw). Finally this type of study is only(unique) in his design since adult population will be evaluated in Mexico.

This study will allow:

1. To evaluate and to compare the experimental vaccine against the virus of the pandemic influenza To (H1N1) produced by Sanofi with the seasonal trivalent vaccine against the influenza.
2. To determine the possibility of predicting the level of immunological response in level terms(ends) of antibodies that the Vaccine pandemic Sanofi produces To (H1N1).
3. To determine the possibility of predicting the frequency of adverse reactions attributed to the Vaccine pandemic Sanofi To (H1N1) evaluated in adult Mexican population. The response will be evaluated of seroconversión (I increase in the titles in four times with regard to the level basal), seropositividad (titles(degrees) overhead of 1:40) and titles(degrees) to geometric averages. The patients will be analyzed in the group in which they were randomized (intention of treatment). The information will be tried using the statistical package SPSS, version 10.1.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* 18 to 60 years old
* Resident in study area
* Available during the time of follow-up
* In good state of health
* Laboratory examinations normal in 28 days before the recruitment
* Negative test(proof) to VIH
* Negative test(proof) to surface antigen of hepatitis B (HBsAg)
* Negative test(proof) to virus of hepatitis C

Exclusion Criteria:

* In women, suckling or plans of pregnancy(embarrassment)
* Ingestion of Medicines immunosuppressants
* Receipt of blood products, 120 days before the screening for VIH
* Receipt of immunoglobulin 60 days before the tamizaje for VIH
* Have received alive(vivacious) attenuated vaccines 30 days to the vaccination
* To have received vaccines unactivated (influenza, pneumococcus or treatment for allergy) in 14 days before the vaccination
* Treatment of latent or active tuberculosis
* History of autoimmune disease or immunodeficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
reactogenicity and safety | day 28, day 56 and day 84

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garcia-Garcia, MD, PhD, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Instituto Nacional de Salud Pública, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Background] Wu B, Huang C, Garcia L, Ponce de Leon A, Osornio JS, Bobadilla-del-Valle M, Ferreira L, Canizales S, Small P, Kato-Maeda M, Krensky AM, Clayberger C. Unique gene expression profiles in infants vaccinated with different strains of Mycobacterium bovis bacille Calmette-Guerin. Infect Immun. 2007 Jul;75(7):3658-64. doi: 10.1128/IAI.00244-07. Epub 2007 May 14. PMID 17502394
- [Background] Wong-Chew RM, Islas-Romero R, Garcia-Garcia Mde L, Beeler JA, Audet S, Santos-Preciado JI, Gans H, Lew-Yasukawa L, Maldonado YA, Arvin AM, Valdespino-Gomez JL. Immunogenicity of aerosol measles vaccine given as the primary measles immunization to nine-month-old Mexican children. Vaccine. 2006 Jan 30;24(5):683-90. doi: 10.1016/j.vaccine.2005.08.045. Epub 2005 Aug 24. PMID 16154241
- [Background] Wong-Chew RM, Islas-Romero R, Garcia-Garcia Mde L, Beeler JA, Audet S, Santos-Preciado JI, Gans H, Lew-Yasukawa L, Maldonado YA, Arvin AM, Valdespino-Gomez JL. Induction of cellular and humoral immunity after aerosol or subcutaneous administration of Edmonston-Zagreb measles vaccine as a primary dose to 12-month-old children. J Infect Dis. 2004 Jan 15;189(2):254-7. doi: 10.1086/380565. Epub 2004 Jan 5. PMID 14722890
- See also: Laboratories of reactives and biologics in Mexico — http://www.birmex.gob.mx/
- See also: OFFICE RESPONSIBLE FOR THE CONTROL OF VACCINATION IN MEXICO — http://www.censia.salud.gob.mx